CLINICAL TRIAL: NCT04125966
Title: NT-proBNP Measurements to Rule-out Heart Failure Among Patients With Atrial Fibrillation: A Prospective Clinical Study
Acronym: ProAF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Randers Regional Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 69531
Record Dates: First submitted 2019-10-04; First posted 2019-10-14 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Atrial Fibrillation; Heart Failure
Keywords: NT-proBNP; Atrial Fibrillation; Heart Failure
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Lithium-heparin blood samples for analysis of NT-proBNP.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate N-terminal pro brain natriuretic peptide (NT-proBNP) as a biomarker to rule out heart failure in patients with atrial fibrillation. Atrial fibrillation and heart failure often co-exist. Heart failure is important to identify, as part of the medical treatment for patients with atrial fibrillation can be fatal if the patient has concomitant heart failure. Performing an echocardiography is considered "gold standard" for assessing cardiac function but echocardiography may not always be readily available during acute hospitalization. The cardiac biomarker NT-proBNP can be used to rule out acute heart failure in patients with sinus rhythm. However, atrial fibrillation affects levels of NT-proBNP in the blood and it is therefore unknown, how the biomarker performs in atrial fibrillation patients.

DETAILED DESCRIPTION:
Background and hypothesis:

Atrial fibrillation is the most common cardiac arrhythmia with a prevalence of approximately 2% in the general population and even higher among elderlies. Atrial fibrillation is associated with an increased morbidity, mortality and risk of heart failure. Patients with atrial fibrillation are at risk of developing tachycardia-induced cardiomyopathy. Furthermore, heart failure of any other cause and atrial fibrillation often co-exist and these patients are at high risk of adverse outcomes and hospitalization. Therefore, early identification of heart failure among patients with atrial fibrillation is important in order to initiate the optimal treatment strategy. However, as recent onset atrial fibrillation and heart failure may present with similar symptoms, excluding heart failure in atrial fibrillation patients is a clinical challenge. The gold standard for evaluating heart failure is echocardiography. However, the access to echocardiographic evaluation may be limited in some hospitals receiving patients with atrial fibrillation. In situations where acute heart failure cannot be ruled-out, clinicians may choose to prescribe digoxin instead of e.g. beta blockers that are preferred for heart rate control. Digoxin is associated with a substantially higher mortality in large cohorts and is not recommended as a first line treatment. Methods other than echocardiography to rule-out heart failure in patients with atrial fibrillation is therefore warranted.

N-terminal pro-brain natriuretic peptide (NT-proBNP) is an established biomarker in identifying and determining long-term prognosis of heart failure in the general population. However, levels of NT-proBNP are known to be higher in atrial fibrillation patients, regardless of underlying structural heart disease.Therefore, it is not possible to rule-out heart failure in patients presenting to the Emergency Department with new-onset atrial fibrillation using existing algorithms for NT-proBNP and heart failure. Accordingly, the aim of this study is to prospectively measure NT-proBNP in atrial fibrillation patients to identify a NT-proBNP threshold making heart failure unlikely.

Perspectives: This study will evaluate if NT-proBNP may be feasible to rule-out heart failure in patients presenting with atrial fibrillation without the use of echocardiography. Early rule-out of heart failure will allow the use of more safe medication for rate control e.g. beta-blockers instead of digoxin.

ELIGIBILITY:
Inclusion Criteria:

* Admission to hospital with atrial fibrillation
* On-going atrial fibrillation documented on an ECG

Exclusion Criteria:

* <18 years
* Other arrhythmias than atrial fibrillation
* Hemodynamically unstable
* Terminal renal failure (in dialysis)
* Pregnancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to the Emergency Department with atrial fibrillation.
Sampling Method: Non-Probability Sample
Enrollment: 403 (Estimated)
Dates: Start 2019-11-11 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of NT-proBNP for ruling out heart failure in atrial fibrillation patients | 0-48 hours after admission to hospital
  The negative predictive value (NPV) of NT-proBNP for ruling out heart failure in atrial fibrillation patients

SECONDARY OUTCOMES:
Overall diagnostic performance of NT-proBNP in detecting heart failure among atrial fibrillation patients | 0-48 hours after admission to hospital
  Sensitivity, specificity and the positive predictive value (PPV)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Løfgren, Professor, MD, PhD, FESC, FAHA, Principal Investigator — Randers Regional Hospital
Locations (1):
- Randers Regional Hospital, Randers, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zoni-Berisso M, Lercari F, Carazza T, Domenicucci S. Epidemiology of atrial fibrillation: European perspective. Clin Epidemiol. 2014 Jun 16;6:213-20. doi: 10.2147/CLEP.S47385. eCollection 2014. PMID 24966695
- [Background] Wang TJ, Larson MG, Levy D, Vasan RS, Leip EP, Wolf PA, D'Agostino RB, Murabito JM, Kannel WB, Benjamin EJ. Temporal relations of atrial fibrillation and congestive heart failure and their joint influence on mortality: the Framingham Heart Study. Circulation. 2003 Jun 17;107(23):2920-5. doi: 10.1161/01.CIR.0000072767.89944.6E. Epub 2003 May 27. PMID 12771006
- [Background] Abualnaja S, Podder M, Hernandez AF, McMurray JJ, Starling RC, O'Connor CM, Califf RM, Armstrong PW, Ezekowitz JA. Acute Heart Failure and Atrial Fibrillation: Insights From the Acute Study of Clinical Effectiveness of Nesiritide in Decompensated Heart Failure (ASCEND-HF) Trial. J Am Heart Assoc. 2015 Aug 24;4(8):e002092. doi: 10.1161/JAHA.115.002092. PMID 26304935
- [Background] McManus DD, Saczynski JS, Lessard D, Kinno M, Pidikiti R, Esa N, Harrington J, Goldberg RJ. Recent trends in the incidence, treatment, and prognosis of patients with heart failure and atrial fibrillation (the Worcester Heart Failure Study). Am J Cardiol. 2013 May 15;111(10):1460-5. doi: 10.1016/j.amjcard.2013.01.298. PMID 23465093
- [Background] Benza RL, Tallaj JA, Felker GM, Zabel KM, Kao W, Bourge RC, Pearce D, Leimberger JD, Borzak S, O'connor CM, Gheorghiade M; OPTIME-CHF Investigators. The impact of arrhythmias in acute heart failure. J Card Fail. 2004 Aug;10(4):279-84. doi: 10.1016/j.cardfail.2003.12.007. PMID 15309692
- [Background] Mountantonakis SE, Grau-Sepulveda MV, Bhatt DL, Hernandez AF, Peterson ED, Fonarow GC. Presence of atrial fibrillation is independently associated with adverse outcomes in patients hospitalized with heart failure: an analysis of get with the guidelines-heart failure. Circ Heart Fail. 2012 Mar 1;5(2):191-201. doi: 10.1161/CIRCHEARTFAILURE.111.965681. Epub 2012 Feb 23. PMID 22361078
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JG, Coats AJ, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GM, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; Authors/Task Force Members; Document Reviewers. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2016 Aug;18(8):891-975. doi: 10.1002/ejhf.592. Epub 2016 May 20. No abstract available. PMID 27207191
- [Background] Bavishi C, Khan AR, Ather S. Digoxin in patients with atrial fibrillation and heart failure: A meta-analysis. Int J Cardiol. 2015 Jun 1;188:99-101. doi: 10.1016/j.ijcard.2015.04.031. Epub 2015 Apr 6. No abstract available. PMID 25900519
- [Background] Turakhia MP, Santangeli P, Winkelmayer WC, Xu X, Ullal AJ, Than CT, Schmitt S, Holmes TH, Frayne SM, Phibbs CS, Yang F, Hoang DD, Ho PM, Heidenreich PA. Increased mortality associated with digoxin in contemporary patients with atrial fibrillation: findings from the TREAT-AF study. J Am Coll Cardiol. 2014 Aug 19;64(7):660-8. doi: 10.1016/j.jacc.2014.03.060. PMID 25125296
- [Background] Chao TF, Liu CJ, Chen SJ, Wang KL, Lin YJ, Chang SL, Lo LW, Hu YF, Tuan TC, Chen TJ, Chiang CE, Chen SA. Does digoxin increase the risk of ischemic stroke and mortality in atrial fibrillation? A nationwide population-based cohort study. Can J Cardiol. 2014 Oct;30(10):1190-5. doi: 10.1016/j.cjca.2014.05.009. Epub 2014 May 14. PMID 25262860
- [Background] Hildebrandt P, Collinson PO, Doughty RN, Fuat A, Gaze DC, Gustafsson F, Januzzi J, Rosenberg J, Senior R, Richards M. Age-dependent values of N-terminal pro-B-type natriuretic peptide are superior to a single cut-point for ruling out suspected systolic dysfunction in primary care. Eur Heart J. 2010 Aug;31(15):1881-9. doi: 10.1093/eurheartj/ehq163. Epub 2010 Jun 2. PMID 20519241
- [Background] Maisel AS, Krishnaswamy P, Nowak RM, McCord J, Hollander JE, Duc P, Omland T, Storrow AB, Abraham WT, Wu AH, Clopton P, Steg PG, Westheim A, Knudsen CW, Perez A, Kazanegra R, Herrmann HC, McCullough PA; Breathing Not Properly Multinational Study Investigators. Rapid measurement of B-type natriuretic peptide in the emergency diagnosis of heart failure. N Engl J Med. 2002 Jul 18;347(3):161-7. doi: 10.1056/NEJMoa020233. PMID 12124404
- [Background] Januzzi JL Jr, Chen-Tournoux AA, Christenson RH, Doros G, Hollander JE, Levy PD, Nagurney JT, Nowak RM, Pang PS, Patel D, Peacock WF, Rivers EJ, Walters EL, Gaggin HK; ICON-RELOADED Investigators. N-Terminal Pro-B-Type Natriuretic Peptide in the Emergency Department: The ICON-RELOADED Study. J Am Coll Cardiol. 2018 Mar 20;71(11):1191-1200. doi: 10.1016/j.jacc.2018.01.021. PMID 29544601
- [Background] Januzzi JL Jr, Camargo CA, Anwaruddin S, Baggish AL, Chen AA, Krauser DG, Tung R, Cameron R, Nagurney JT, Chae CU, Lloyd-Jones DM, Brown DF, Foran-Melanson S, Sluss PM, Lee-Lewandrowski E, Lewandrowski KB. The N-terminal Pro-BNP investigation of dyspnea in the emergency department (PRIDE) study. Am J Cardiol. 2005 Apr 15;95(8):948-54. doi: 10.1016/j.amjcard.2004.12.032. PMID 15820160
- [Background] Jin M, Wei S, Gao R, Wang K, Xu X, Yao W, Zhang H, Zhou Y, Xu D, Zhou F, Li X. Predictors of Long-Term Mortality in Patients With Acute Heart Failure. Int Heart J. 2017 May 31;58(3):409-415. doi: 10.1536/ihj.16-219. Epub 2017 May 12. PMID 28496020
- [Background] Knudsen CW, Omland T, Clopton P, Westheim A, Wu AH, Duc P, McCord J, Nowak RM, Hollander JE, Storrow AB, Abraham WT, McCullough PA, Maisel A. Impact of atrial fibrillation on the diagnostic performance of B-type natriuretic peptide concentration in dyspneic patients: an analysis from the breathing not properly multinational study. J Am Coll Cardiol. 2005 Sep 6;46(5):838-44. doi: 10.1016/j.jacc.2005.05.057. PMID 16139134
- [Background] Lauridsen KG, Schmidt AS, Adelborg K, Bach L, Hornung N, Jepsen SM, Deakin CD, Rickers H, Lofgren B. Effects of hyperoxia on myocardial injury following cardioversion-A randomized clinical trial. Am Heart J. 2018 Feb;196:97-104. doi: 10.1016/j.ahj.2017.10.006. Epub 2017 Oct 14. PMID 29421020
- [Derived] Budolfsen C, Schmidt AS, Lauridsen KG, Hoeks CB, Waziri F, Poulsen CB, Riis DN, Rickers H, Lofgren B. NT-proBNP cut-off value for ruling out heart failure in atrial fibrillation patients - A prospective clinical study. Am J Emerg Med. 2023 Sep;71:18-24. doi: 10.1016/j.ajem.2023.05.041. Epub 2023 Jun 7. PMID 37320999